CLINICAL TRIAL: NCT06001775
Title: Embedded Clinical Trial of Patient Priorities Care Among Persons Living With Mild Cognitive Impairment and Dementia
Brief Title: Patient Priorities Care Among Persons Living With Mild Cognitive Impairment and Dementia
Acronym: IN-TX-PPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jennifer L Carnahan, Research Scientist, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FY22_Pilot1_Carnahan; 15345 (Other: Indiana University Institutional Review Board); Pro00063400 (Other: Advarra (CIRBI) External Institutional Review Board); U54AG063546 (NIH)
Record Dates: First submitted 2023-08-07; First posted 2023-08-21 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Dementia; Mild Cognitive Impairment
Keywords: dementia; mild cognitive impairment; patient priorities care
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Priorities Care Eligible Persons Living With Dementia and Mild Cognitive Impairment (Experimental): Patients (and their care partners when available) will receive a packet of information about Patient Priorities Care, and when feasible, a trained facilitator(s) will initiate a Patient Priorities Care conversation with the patient or patient care partner dyad. This conversation will be documented in the Electronic Health Record.
  Interventions: Behavioral: Patient Priorities Care

INTERVENTIONS:
Behavioral: Patient Priorities Care — According to patientprioritiescare.org a Patient Priorities Care conversation helps to align healthcare decision-making and care by all clinicians with patients' own health priorities. Patient Priorities Care involves not only the health outcome goals that patients want to achieve, but also their preferences for healthcare.

SUMMARY:
The goal of this pragmatic, embedded clinical trial is to analyze the implementation of Patient Priorities Care in primary care and geriatrics clinics with patients living with dementia or mild cognitive impairment. This study aims are:

* demonstrate the feasibility of using the electronic health record to identify a diverse cohort of eligible patient and patient-care partner dyads who will engage in a Patient Priorities Care conversation with a trained facilitator.
* demonstrate feasibility of pragmatically assessing clinical outcomes using the electronic health record, including a) number of days at home, b) total medications, and c) new referrals to specialist physicians.
* examine key feasibility measures across racial, ethnic, and socioeconomic subgroups.

Participants will receive a packet of information about Patient Priorities Care from their primary care clinic, in advance of their next upcoming clinic appointment. Individuals who receive a packet will have the opportunity to engage in a conversation about what matters most to them and what their priorities are, with trained facilitators at the clinic.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria

Patients must meet all of the following criteria to participate in this study:

* 40 years or older

  * English-speaking at both Indiana sites or English and/or Spanish speaking at the University of Texas site
  * Receiving care with a participating physician
  * Has a scheduled outpatient care visit within 1-2 months (60 days)
  * Individual has a diagnosis of MCI or dementia

Definition: To identify individuals with dementia and MCI, we will use two or more instances of use of an ICD-10 code for either diagnosis in the EHR within 24 months. Typically, we would include instances of these billing codes within a year of each other but, due to the COVID-19 pandemic, recognize that there may be less frequent clinical visits and less robust billing. Diagnostic codes include:

• F01.50, F01.51, F02.80, F02.81, F03.90, G30.0, G30.1, G30.8, G30.9, G31.01, G31.09, G31.1, G31.2, F41.81, G31.84 and F03.91.

Care Partner Inclusion Criteria

Care partners must meet all of the following criteria to participate in the study:

* 18 years or older
* English-speaking at both Indiana sites or English and/or Spanish speaking at the University of Texas site

A note about inclusion of care partners: Clinician determination of a patient's capacity to participate in a visit independently is part of a pragmatic approach. This means that clinic staff will determine when a care partner is needed. Generally, we act under the assumption that patients who require a care partner will have already included them in previous visits and/or provider communications (and we anticipate that this will be documented in the EHR), whereas patients who attend clinic visits independently and have no documentation indicating the involvement of a care partner in their medical decisions, or a need for one, will be determined to have the capacity to also participate in a PPC visit.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from the study:

* Is not community-dwelling- e.g. lives in a nursing home
* Is enrolled in hospice
* Individuals who decline to receive the PPC intervention (i.e. decline to have the PPC conversation) will be excluded from the study.

  * Note that declining to receive the PPC intervention will in no way impact the care that patients receive now or in the future.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Documentation of PPC discussion | Baseline
  Review of the electronic health record will be used to assess for the presence of documentation of patient priorities care for each enrolled patient.

SECONDARY OUTCOMES:
Identification of a care partner | Baseline and up to 2 months post baseline
  Identification of a care partner for 50% of eligible persons living with dementia and mild cognitive impairment. Care partners will be identified based on information provided by the patient, the electronic health record, and the clinical team.
Acceptability | Baseline and up to 2 months post baseline
  Acceptability will be assessed using Sekhon's Theoretical Framework of Acceptability (TFA) to qualitatively assess acceptability, which includes meeting definitions outlined within the framework, represented by seven component constructs: affective attitude, burden, perceived effectiveness, ethicality, intervention coherence, opportunity costs, and self-efficacy.
Appropriateness | Baseline and up to 2 months post baseline
  Appropriateness will be assessed via qualitative exit interviews with patients, care partners, and clinicians.
Feasibility of the intervention | Baseline and up to 2 months post baseline
  Feasibility will be assessed qualitatively using the description provided by Proctor et al as a guide.
Fidelity to the intervention | Baseline and up to 2 months post baseline
  Fidelity will be assessed when select charts are reviewed for adherence to the protocol.
Potential for future adoption of Patient Priorities Care intervention | Baseline and up to 2 months post baseline
  Assessment of potential for future adoption of the intervention will be conducted via qualitative exit interviews with patients, care partners, and clinicians.
Number of patient days at home | 2 months pre and 2 months post baseline
  Review of the electronic health record will be used to assess for hospital visits, emergency room visits, or nursing home admissions. Number of patient days at home will be further evaluated across racial, ethnic, and socioeconomic subgroups to detect any differences.
Number of total medications | 2 months pre and 2 months post baseline
  Review of the electronic health record will be used to assess the medication list total at 2 months pre and post baseline. Number of total medications will be further evaluated across racial, ethnic, and socioeconomic subgroups to detect any differences.
Number of new referrals to specialist physicians | 2 months pre and 2 months post baseline
  Review of the electronic health record to identify the number of referrals to specialists at 2 months pre and post baseline. Number of new referrals to specialist physicians will be further evaluated across racial, ethnic, and socioeconomic subgroups to detect any differences.
Number of patients across racial, ethnic, and socioeconomic subgroups with documentation of Patient Priorities Care discussion in the electronic health record | 2 months pre and 2 months post baseline
  Evaluation will occur using a previously established natural language processing model to identify patient medical records when a Patient Priorities Care discussion is recorded.
Acceptability across racial, ethnic, and socioeconomic subgroups. | Baseline and up to 2 months post baseline
  Acceptability effects will be further evaluated across racial, ethnic, and socioeconomic subgroups. We will utilize Sekhon et al's Theoretical Framework of Acceptability (TFA) to qualitatively assess acceptability, which includes meeting definitions outlined within the framework, represented by seven component constructs: affective attitude, burden, perceived effectiveness, ethicality, intervention coherence, opportunity costs, and self-efficacy.
Number of Patients with Social Factors Indicated in the Electronic Health Record | Baseline and up to 2 months post baseline
  Established algorithms for detecting social factors that may influence patient care priorities, such as housing instability, financial insecurity, or transportation concerns will be deployed. These algorithms have been previously created and validated across the care spectrum and will be deployed at the primary site in current form on the established natural language processing platform at Regenstrief Institute. Similar data will be manually extracted using keywords from the primary site for the secondary site. All available clinical notes for the recruited cohort will be annotated by the software as either positive or negative for the social factors. This can then be incorporated into analyses.

OTHER OUTCOMES:
Number of Enrolled Eligible Dyads across racial, ethnic and socioeconomic subgroups | 2 months pre and 2 months post baseline
  Number of eligible dyads enrolled across racial, ethnic and socioeconomic subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Carnahan, MD, Principal Investigator — Regenstrief Institute, Inc.
Locations (3):
- United States (3):
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University Health Connected Care, Indianapolis, Indiana
  - University of Texas Health- Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Since this study is a pragmatic trial in a clinical environment, the majority of our outcomes will be determined via data that is already held in the EHR. Therefore a plan for sharing IPD seems unnecessary.

REFERENCES:
- See also: Patient Priorities Care homepage — http://patientprioritiescare.org